CLINICAL TRIAL: NCT06160479
Title: The Incidence of Hypocalcemia in Pregnant Women at Siriraj Hospital
Acronym: HypoCal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Tachjaree Panchalee, Assistant Professor Tachjaree Panchalee, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Si 1003/2021
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Hypocalcemia in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal calcium level with no receiving calcium supplement (No Intervention): Pregnant women with normal calcium level in the first half of pregnancy do not receive calcium supplement.
- Normal calcium level with receiving calcium supplement 1g/day (Experimental): Pregnant women with normal calcium level in the first half of pregnancy receive calcium supplement 1g/day.
  Interventions: Drug: Calcium supplement
- Hypocalcemia with receiving calcium supplement 1g/day (Experimental): Pregnant women with hypocalcemia in the first half of pregnancy receive calcium supplement 1g/day.
  Interventions: Drug: Calcium supplement
- Hypocalcemia level with receiving calcium supplement 2g/day (Experimental): Pregnant women with hypocalcemia in the first half of pregnancy receive calcium supplement 2g/day.
  Interventions: Drug: Calcium supplement

INTERVENTIONS:
Drug: Calcium supplement — Different amount of calcium supplement in pregnancy
  Arms: Hypocalcemia level with receiving calcium supplement 2g/day; Hypocalcemia with receiving calcium supplement 1g/day; Normal calcium level with receiving calcium supplement 1g/day

SUMMARY:
Calcium is an essential element for fundamental physiological functions and during pregnancy. However, higher calcium intake can induce constipation, flatulence, nausea, or kidney stones. This study aims to evaluate the incidence of hypocalcemia among pregnant women in the first half of pregnancy in Thailand. Also, Comparison of calcium level in pregnant women in the third trimester who received and not received calcium during pregnancy.

DETAILED DESCRIPTION:
The primary outcome is the incidence of hypocalcemia among pregnant women in the first half of pregnancy. This study also has secondary objectives. The one is associating factors with calcium level. After getting the results of maternal calcium level, the normal calcium level group will be divided into 2 groups for receiving calcium 1 g/day and no receiving calcium supplement. Another with hypocalcemia group will be decided into 2 groups for receiving calcium 1 g/day and 2 g/day. The calcium level was collected again in the third trimester.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who attend antenatal care clinic in Siriraj Hospital
* Pregnant women with gestation less than 20 weeks of gestation
* Singleton pregnancy

Exclusion Criteria:

* Pregnant women who has underlying diseases including liver disease and vitamin D deficiency
* Pregnant women are malnutrition patients
* Pregnant women who receive calcium supplement before enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypocalcemia in pregnant women at Siriraj Hospital | 1.5 year
  The incidence of hypocalcemia in pregnant women in the first half of pregnancy. Material blood will be taken for calcium level. The hypocalcemia is defined as total calcium level less than 8.5 mg/dl.

SECONDARY OUTCOMES:
The demographic and pregnant factors are associating with maternal calcium level in the first half of pregnancy assessed by the questionnaire and scrupulous chart review | 1.5 year
  The different characteristics between normal calcium and hypocalcemia group in the first half of pregnancy will be studied. The data will be received by interviewing the patients, answering the questionnaire and scrupulous chart review; including age, education, occupations, income, marital status, food and nutrition status, previous pregnancy outcomes, family history, mode of conception in this pregnancy, gestational age of blood drawing, caffeine intake, smoking, and maternal hematocrit.
The calcium level in pregnant women in the third trimester | 2 year
  Comparison of maternal serum calcium level in pregnant women in the third trimester between who receive and do not receive calcium supplement. In the normal calcium level group, pregnant women will be divided into 2 groups: receiving CaCO3 1 g/day and no receiving. In the hypocalcemia group, pregnant women will be divided into 2 groups: receiving CaCO3 1g/day and 2g/day. Maternal blood taking for serum calcium level will be done in all participants. Comparison of maternal calcium level between groups will be reported. Statistical analysis will be used t-test and p-value is less than 0.5.

CONTACTS AND LOCATIONS:
Overall Officials: Tachjaree Panchalee, MD, Study Director — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand